CLINICAL TRIAL: NCT04884334
Title: Data Collection on the Treatment of Gastrointestinal Leakage by the Use of Combination of Covered Nitinol Stent and Negative Pressure Wound Treatment
Brief Title: VAC-Stent Registry
Status: Recruiting | Type: Observational
Sponsor: Markus M. Heiss (Other)
Collaborators: VAC Stent GmbH (Unknown); Möller Medical GmbH (Unknown); MicroTech Europe GmbH (Unknown); University of Witten/Herdecke (Other)
Responsible Party: Sponsor-Investigator, Markus M. Heiss, Prof Dr, University of Witten/Herdecke
Organization: University of Witten/Herdecke (Other)
Other Study IDs: VAC-Stent Registry
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Perforation of the Oesophagus; Perforation of the Colon
Keywords: Perforation Oesophagus; Oesophageal Anastomotic Leak; endoscopic vacuum therapy; Perforation Colon
MeSH Terms: conditions — Esophageal Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VAC-Stent® treatment: spontaneous, iatrogenic or postoperative leakage of the oesophagus or colon
  Interventions: Device: VAC-Stent®

INTERVENTIONS:
Device: VAC-Stent® — treatment with the VAC-Stent®

SUMMARY:
This registry is intended to collect data on quality assurance and use of the VAC-Stent® and thus verify the suitability of the VAC-Stent® for sealing leakages in the oesophagus or colon. Furthermore, the safety and efficacy of the VAC-Stent® shall be proven.

DETAILED DESCRIPTION:
For this registry, quality assurance data will be prospectively collected from all patients who receive the VAC-Stent®. The VAC-Stent® combines a vacuum sponge, which lies intraluminal and conditions the wound, with a covered stent, which seals the sponge from the lumen and thus ensures passage. Due to its design, the new medical device VAC-Stent® offers a solution for the most important problems of the covered stent, the stent migration and the lack of drainage function, as well as for those of the endoluminal vacuum sponge, the blockage of the gastrointestinal lumen and the difficult application. The VAC-Stent® is the technical advancement for all indications of the covered stent and for the indication of the endoluminal vacuum sponge, so that a very good effectiveness with reduced complications can be expected for these clinical situations.

The VAC-Stent® therefore offers the prospect of an innovative further development in the endoscopic treatment of leaks in the gastrointestinal tract, without any new and unknown risks being associated with it.

The primary aim of this registry is to collect data on the quality assurance and application of the VAC-Stent® and thus to evaluate the suitability of the VAC-Stent® for sealing leaks in the oesophagus or colon. In addition, the safety and efficacy of the VAC-Stent® will be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* treatment with the VAC-Stent®

Exclusion Criteria:

- accommodation in an institution under court or administrative order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spontaneous, iatrogenic or postoperative leakages in the oesophagus or colon
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Successful treatment of the leakage with the VAC-Stent® | up to 6 months

SECONDARY OUTCOMES:
Rate of morphological healing of the insufficiency | approximately 4 weeks after end of treatment
Number of Participants with complications | approximately 4 weeks after end of treatment

CONTACTS AND LOCATIONS:
Locations (14):
- Germany (14):
  - Charité, Berlin
  - Sana Klinikum Lichtenberg, Berlin
  - St. Josef-Hospital, Bochum
  - Johanniter Krankenhaus Bonn, Bonn
  - Ameos Klinikum Am Bürgerpark, Bremerhaven
  - Allgemeines Krankenhaus Celle, Celle
  - Visceral, Tumour, Vascular and Transplant Surgery, Cologne Merheim Hospital, Cologne
  - Städtisches Klinikum Dresden, Dresden
  - Uniklinik Düsseldorf, Düsseldorf
  - KRH Klinikum Siloah, Hanover
  - Nils Stensen Kliniken, Marienhospital Osnabrück, Osnabrück
  - Caritas Klinikum Saarbrücken - St. Theresia, Saarbrücken
  - Uniklinik Tübingen, Tübingen
  - Asklepios Paulinen Klinik Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heiss MM, Lange J, Knievel J, Yohannes A, Hugle U, Dormann AJ, Eisenberger CF. Treatment of anastomotic leak in colorectal surgery by endoluminal vacuum therapy with the VACStent avoiding a stoma - a pilot study. Langenbecks Arch Surg. 2024 Jul 31;409(1):234. doi: 10.1007/s00423-024-03426-5. PMID 39083099
- [Derived] Lange J, Knievel J, Wichmann D, Kahler G, Wiedbrauck F, Hellmich T, Kandler M, Bernhardt J, Scholz D, Beyna T, Hausmann J, Wedi E, Ellrichmann M, Hugle U, Dormann AJ, Eisenberger CF, Heiss MM. Clinical implantation of 92 VACStents in the upper gastrointestinal tract of 50 patients-applicability and safety analysis of an innovative endoscopic concept. Front Surg. 2023 May 5;10:1182094. doi: 10.3389/fsurg.2023.1182094. eCollection 2023. PMID 37215348